CLINICAL TRIAL: NCT04546061
Title: Project Uplift: Substance Use and Mental Health Treatment for Young Sexual and Gender Minorities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103883; 1H79TI081999 (Other Grant/Funding Number: SAMHSA)
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Substance Use; Mental Health
Keywords: Sexual and Gender Minorities; Substance Use and Mental Health Treatment; Mental Health; Substance Use; Minority Stress; Young Adults; Intensive Case Management; Peer Support
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Project Uplift Intervention (Experimental): A 6-month long intervention for young adult sexual and gender minorities, ages 18-35.
  Interventions: Behavioral: Project Uplift

INTERVENTIONS:
Behavioral: Project Uplift — Substance use and mental health treatment for young sexual and gender minorities in Durham and Charlotte, NC in conjunction with intensive wraparound services that address factors that influence substance use and mental health among this population.

SUMMARY:
This study provides substance use and mental health treatment for young sexual and gender minority adults in Durham and Charlotte, NC and seeks to provide intensive wraparound services that address factors that influence substance use and mental health among this population such as minority stressors and lack of social support, housing instability, lack of access to affirmative health care, and limited job opportunities.

DETAILED DESCRIPTION:
Project Uplift provides evidenced-based substance use and mental health treatment, intensive case management, and peer support services for sexual and gender minorities, ages 18-35. The program is based in two metropolitan areas in North Carolina, Durham and Charlotte, and will offer services for approximately 80 sexual and gender minority young adults. Survey data collected from participants at baseline and at the end of the 6-month program will be used to evaluate the effectiveness the comprehensive care program.

ELIGIBILITY:
Inclusion Criteria: 1) age 18-35; 2) substance use in the last 90 days; 3) self-identify as a sexual and/or gender minority; 4) reside in the Durham or Charlotte geographic areas including neighboring counties

Exclusion Criteria: 1) inability to speak and read English

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Change in substance use from baseline to 6-month follow-up | Baseline and 6-months
  Addiction Severity Index collected via a computer assisted self-interviewing survey
Change in mental health status from baseline to 6-month follow-up | Baseline and 6-months
  Brief Symptom Inventory collected via a computer assisted self-interviewing survey

CONTACTS AND LOCATIONS:
Overall Officials: Sara H LeGrand, PhD, Principal Investigator — Duke University; Susan Reif, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Mecklenburg County Community Support Services, Charlotte, North Carolina
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT04546061/ICF_000.pdf